CLINICAL TRIAL: NCT02078713
Title: Patient-Centered Support for Contraceptive Decision-Making: A Cluster Randomized Controlled Trial of a Contraceptive Decision Support Tool
Brief Title: Patient-Centered Support for Contraceptive Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CE-1304-6874
Record Dates: First submitted 2014-02-25; First posted 2014-03-05 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-04

CONDITIONS: Contraception; Contraceptive Behavior
Keywords: contraception; patient decision support; patient decision aid; shared decision making; Decision Making, Shared; Patient-Centered Outcomes Research
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contraceptive Decision Support Tool (Experimental): Patients whose contraceptive counseling visits are scheduled with providers randomized to this arm will use the intervention immediately before their visit and bring the generated printout to their visit. Providers randomized to this arm will be free to integrate the tool and printout into their contraceptive counseling however they see fit.
  Interventions: Behavioral: Contraceptive Decision Support Tool
- Usual Care (Control) (No Intervention): Patients in this arm will receive usual family planning care.

INTERVENTIONS:
Behavioral: Contraceptive Decision Support Tool — The decision support tool:
  * Provides an educational session about different aspects of contraception
  * Elicits patient preferences about different aspects of contraception
  * Identifies potential contraindications to certain contraceptive methods
  * Allows the patient to view details about and compare available contraceptive methods
  * Suggests methods most appropriate based on the patient's preferences
  * Collects questions the patient may have for her provider
  * Generates a printout the patient can bring to her contraceptive counseling visit
  Arms: Contraceptive Decision Support Tool

SUMMARY:
The investigators have designed a tablet-based decision support tool to help women learn more about their birth control options and support them in choosing a method they are happy with. The investigators will test whether the decision support tool helps women choose a birth control method they can continue using successfully by having some women use the tool before their birth control-related visit to a health care provider, and some women not use the tool before their visit. The investigators will then follow up with all the women at four months and seven months after their visit to see if they are still using the birth control method they chose at the visit and how happy they are with the method.

Hypotheses:

1. Women who use the contraceptive decision support tool will be more likely to continue using their chosen method at 4 and 7 months follow-up, compared to women who receive usual care.
2. The contraceptive decision support tool will increase women's knowledge, choice of, and use of highly effective reversible contraception, compared to usual care.
3. The contraceptive decision support tool will decrease decision conflict, compared to usual care.
4. The contraceptive decision support tool will increase patient satisfaction with the clinic visit and with their method, compared to usual care.
5. Women who use the contraceptive decision support tool will have fewer unintended pregnancies during the follow-up period, compared to women who received usual care.
6. The contraceptive decision support tool will increase shared patient-provider decision making in contraceptive counseling visits, compared to usual care.
7. The contraceptive decision support tool will decrease provider frustration when providing contraceptive counseling and increase provider job satisfaction.
8. Women using the tool will be more likely to report use of any moderately or highly effective method of contraception at 4 and 7 months follow-up, compared to women not using the tool.

DETAILED DESCRIPTION:
The impacts of unintended pregnancy include adverse maternal and infant outcomes for women who continue their pregnancies, with higher rates of infant low birth weight, infant mortality, and maternal mortality and morbidity for these pregnancies as compared to planned pregnancies. In addition, children resulting from unplanned pregnancies have been found to be more likely to experience developmental delay.

Over the past several decades, the proportion of unintended pregnancy in the United States has remained stubbornly high at approximately 50%. Each year, one in 20 women of reproductive age experiences an unintended pregnancy, and it is estimated that over half of women will have an unintended pregnancy in their lifetime. This high rate of unintended pregnancy in the United States places a heavy burden on both women and the health care system. A disproportionate amount of this burden is experienced by minority women and women of lower socioeconomic status. Given the high rate of unintended pregnancies in this country, interventions designed to help women achieve their fertility goals could have a substantial impact on their health outcomes and life course. In addition, identifying strategies that are appropriate for use in high-risk, diverse populations could address disparities in women's ability to plan their pregnancies.

The investigators propose a cluster randomized trial to investigate the effect of an interactive, tablet-based contraceptive decision support tool that women will use immediately prior to their contraceptive counseling visits. The goal of the tool is to facilitate shared decision-making between the woman and her health care provider, with the ultimate goal of helping the woman to choose a contraceptive method that is consistent with her values and preferences, and is therefore best suited to helping her to avoid an unplanned pregnancy. The tool will be available in both English and Spanish.

The investigators will measure the tool's effect on women's contraceptive continuation, as well as on their experience of contraceptive counseling, measured both quantitatively and qualitatively. In addition, the investigators will collect quantitative and qualitative data to determine the impact of the implementation of this tool on the experiences of providers and the clinics in which they work.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Women of reproductive age (15-45)
* Wish to discuss starting or changing a contraceptive method during their visit
* Speak, read, and understand English or Spanish (Note: for the pre- and post-intervention audio recording phases, only patients who can speak, read, and understand English easily will be enrolled.)
* History of sexual activity with men

Providers

* Provide contraceptive counseling in one of the participating clinics
* Plan to remain in job role for at least six months

Clinic staff

* Work at one of the participating clinics
* Had a job that included patient contact, but did not solely consist of family planning counseling at the time of the implementation of the intervention

Exclusion Criteria:

Patients

* Previously enrolled in the study
* Previously used the decision support tool at the Women's Community Clinic in San Francisco
* Are unable to get pregnant
* Appointment reason is for insertion of IUD or contraceptive implant
* Currently pregnant
* Desire pregnancy currently or in the next seven months (Note: The last criterion is designed to ensure we will have limited numbers of women that will discontinue their contraceptive methods during the study due to planning a pregnancy.)

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 786 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - San Francisco City Clinic, San Francisco, California
  - Planned Parenthood San Francisco Health Center, San Francisco, California
  - San Francisco General Hospital Family Planning Clinic, San Francisco, California
  - City College of San Francisco Student Health Services, San Francisco, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holt K, Kimport K, Kuppermann M, Fitzpatrick J, Steinauer J, Dehlendorf C. Patient-provider communication before and after implementation of the contraceptive decision support tool My Birth Control. Patient Educ Couns. 2020 Feb;103(2):315-320. doi: 10.1016/j.pec.2019.09.003. Epub 2019 Sep 4. PMID 31537316
- [Derived] Dehlendorf C, Fitzpatrick J, Fox E, Holt K, Vittinghoff E, Reed R, Campora MP, Sokoloff A, Kuppermann M. Cluster randomized trial of a patient-centered contraceptive decision support tool, My Birth Control. Am J Obstet Gynecol. 2019 Jun;220(6):565.e1-565.e12. doi: 10.1016/j.ajog.2019.02.015. Epub 2019 Feb 11. PMID 30763545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female patients were approached to participate in the study before appointments at four San Francisco Bay Area clinics between December 2014 and March 2016.
  Patients are grouped in cluster by provider. Providers of family planning care at the four clinics were approached to participate in the study in October to December 2014.
Pre-assignment Details: A total of 2,458 patients were approached to participate in the study. Of these, 1,700 were excluded before assignment (1,642 due to ineligibility, 58 refusals), and 758 enrolled.
  A total of 36 providers were approached to participate. Eight were excluded before assignment (7 due to ineligibility, 1 refusal), and 28 enrolled.
Groups:
- Contraceptive Decision Support Tool Patients: Patients whose contraceptive counseling visits are scheduled with providers randomized to this arm will use the intervention immediately before their visit and bring the generated printout to their visit. Providers randomized to this arm will be free to integrate the tool and printout into their contraceptive counseling however they see fit.
  Contraceptive Decision Support Tool: The decision support tool:
  * Provides an educational session about different aspects of contraception
  * Elicits patient preferences about different aspects of contraception
  * Identifies potential contraindications to certain contraceptive methods
  * Allows the patient to view details about and compare available contraceptive methods
  * Suggests methods most appropriate based on the patient's preferences
  * Collects questions the patient may have for her provider
  * Generates a printout the patient can bring to her contraceptive counseling visit
- Usual Care (Control) Patients: Patients in this arm will receive usual family planning care.
- Contraceptive Decision Support Tool Providers: Family planning providers randomized to use the Contraceptive Decision Support tool with their patients in the study.
- Usual Care (Control) Providers: Family planning providers randomized to deliver usual care to their patient in the study.
Period: Overall Study
Arm/Group | Contraceptive Decision Support Tool Patients | Usual Care (Control) Patients | Contraceptive Decision Support Tool Providers | Usual Care (Control) Providers
Started | 407 | 351 | 15 | 13
Completed | 355 | 290 | 15 | 13
Not Completed | 52 | 61 | 0 | 0
Not completed — Lost to Follow-up | 49 | 55 | 0 | 0
Not completed — Pregnant at baseline | 3 | 5 | 0 | 0
Not completed — Enrolled twice | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 758 patients enrolled in the study. Patients were excluded post-randomization if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1), for a resultant baseline sample of 749 patients.
Groups:
- Contraception Decision Support Tool Providers: Family planning providers randomized to use the Contraceptive Decision Support tool with their patients. Providers were the unit of randomization in this cluster trial
- Usual Care (Control) Providers: Family planning providers randomized to practice usual care with their patients. Providers were the unit of randomization in this cluster trial
- Total: Total of all reporting groups
Arm/Group | Contraceptive Decision Support Tool Patients | Usual Care (Control) Patients | Contraception Decision Support Tool Providers | Usual Care (Control) Providers | Total
Number analyzed (Participants) | 404 | 345 | 15 | 13 | 777
Age, Customized [Count of Participants; unit: Participants] — Population: Patients were excluded if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1).
  Participants
    Age category: 15-19 | 52 | 43 | 0 | 0 | 95
    Age category: 20-24 | 126 | 121 | 2 | 1 | 250
    Age category: 25-29 | 110 | 91 | 2 | 3 | 206
    Age category: 30-34 | 68 | 53 | 1 | 3 | 125
    Age category: 35-39 | 33 | 22 | 2 | 1 | 58
    Age category: 40-45 | 13 | 10 | 4 | 1 | 28
    Age category: Over 45 | 0 | 0 | 4 | 4 | 8
    Age category: Missing | 2 | 5 | 0 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 404 | 345 | 15 | 12 | 776
  Male | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Patients were excluded from analysis if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1).
  Participants
    Race/ethnicity: African American/Black | 46 | 34 | 0 | 0 | 80
    Race/ethnicity: Asian or Pacific Islander | 59 | 62 | 2 | 0 | 123
    Race/ethnicity: Hispanic/Latina | 160 | 128 | 4 | 4 | 296
    Race/ethnicity: White | 86 | 85 | 8 | 9 | 188
    Race/ethnicity: Other | 51 | 32 | 1 | 0 | 84
    Race/ethnicity: Missing | 2 | 4 | 0 | 0 | 6
Language spoken during study participation [Count of Participants; unit: Participants] — Population: Patients were excluded from analysis if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1).
  Participants
    English | 329 | 283 | 15 | 13 | 640
    Spanish | 75 | 62 | 0 | 0 | 137
Parental education [Count of Participants; unit: Participants] — Population: Patients were excluded from analysis if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1).
  These data were not collected from the provider sample.
  Participants
    number analyzed (Participants) | 404 | 345 | 0 | 0 | 749
    8th grade or less | 69 | 50 | 0 | 0 | 119
    Some high school, but did not graduate | 38 | 29 | 0 | 0 | 67
    High school graduate or GED | 81 | 69 | 0 | 0 | 150
    Some college or 2-year degree | 83 | 58 | 0 | 0 | 141
    4-year college graduate or more | 129 | 133 | 0 | 0 | 262
    Missing | 4 | 6 | 0 | 0 | 10
% Federal Poverty Line [Count of Participants; unit: Participants] — Population: Patients were excluded from analysis if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1).
  These data were not collected from the provider sample.
  Participants
    number analyzed (Participants) | 404 | 345 | 0 | 0 | 749
    <100% | 183 | 141 | 0 | 0 | 324
    101-200% | 81 | 79 | 0 | 0 | 160
    >200% | 76 | 65 | 0 | 0 | 141
    Missing | 64 | 60 | 0 | 0 | 124
Parity [Count of Participants; unit: Participants] — Population: Patients were excluded from analysis if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1).
  These data were not collected from the provider sample.
  Participants
    number analyzed (Participants) | 404 | 345 | 0 | 0 | 749
    Nulliparous | 265 | 236 | 0 | 0 | 501
    Parous | 133 | 104 | 0 | 0 | 237
    Missing | 6 | 5 | 0 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Contraceptive Continuation
Description: Whether or not a participant is still using the contraceptive method she selected at baseline.
Time Frame: 4 and 7 months post-enrollment
Population: Analysis was modified intention to treat. In accordance with the statistical analysis plan, patients were excluded from analysis if they were pregnant at baseline (n=8) or enrolled in the study twice (n=1, in which case information from their second enrollment was excluded). Outcome observed in patients only.
Measure: Count of Participants; unit: Participants
Groups:
- Contraceptive Decision Support Tool: Patients whose contraceptive counseling visits are scheduled with providers randomized to this arm will use the intervention immediately before their visit and bring the generated printout to their visit. Providers randomized to this arm will be free to integrate the tool and printout into their contraceptive counseling however they see fit.
  Contraceptive Decision Support Tool: The decision support tool:
  * Provides an educational session about different aspects of contraception
  * Elicits patient preferences about different aspects of contraception
  * Identifies potential contraindications to certain contraceptive methods
  * Allows the patient to view details about and compare available contraceptive methods
  * Suggests methods most appropriate based on the patient's preferences
  * Collects questions the patient may have for her provider
  * Generates a printout the patient can bring to her contraceptive counseling visit
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  7 months post-enrollment: Continuous user of chosen method | 201 | 174
  7 months post-enrollment: Not a continuous user of chosen method | 154 | 118
  7 months post-enrollment: Missing | 49 | 53
  4 months post-enrollment: Continuous user of chosen method | 249 | 228
  4 months post-enrollment: Not a continuous user of chosen method | 115 | 83
  4 months post-enrollment: Missing | 40 | 34
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 7 months post-enrollment; Test type: Superiority; p = 0.46, Regression, Logistic — P-value calculated in multiply imputed dataset; We ran a mixed effect regression model in a multiply imputed dataset, using fixed effects for study site and random effects for provider seen; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.65 to 1.22] — The odds ratio represents the odds of the intervention group in the numerator over the odds of the control group in the denominator
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 4 months post-enrollment; Test type: Superiority; p = 0.16, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.57 to 1.10] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Patient Contraceptive Counseling Satisfaction
Description: Patient-reported score on an 11-item factor analysis-validated measure created by the PI to assess patients' satisfaction with the contraceptive counseling experience. The measure consists of 5-point Likert scale items on which patients evaluate provider performance, with item response options ranging from 1 ("Poor") to 5 ("Excellent"). The score range for the total measure is11-55, with 11 as the worst possible score and 55 as the best possible score for provider performance. Analyzed dichotomously, top score (55) versus all lower scores.
Time Frame: Baseline, post-visit survey
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Top score of 55 | 261 | 194
  Less than top score of 55 | 133 | 143
  Missing | 10 | 8
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p = 0.03, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.03 to 2.05] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Patient Satisfaction With Information Received About Side Effects During Counseling
Description: Patient response to a 5-point Likert scale item about satisfaction with information that their provider gave them about side effects of their chosen methods during their baseline visit (1=completely unsatisfied, 5=completely satisfied). Analyzed dichotomously as top score of 5 versus <5.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool Patients | Usual Care (Control) Patients
Number analyzed (Participants) | 404 | 345
Participants
  Top score of 5, completely satisfied | 325 | 253
  Less than 5 | 64 | 81
  Missing | 15 | 11
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool Patients vs Usual Care (Control) Patients; Test type: Superiority; p = 0.01, Regression, Logistic — P-value calculated in imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.11 to 2.33] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Satisfaction With Visit
Description: Patient report on 5-point Likert scale of satisfaction with baseline visit (1=completely unsatisfied, 5=completely satisfied). Analyzed dichotomously as top score of 5 versus <5.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Completely satisfied | 338 | 282
  Less than completely satisfied | 56 | 54
  Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p = 0.62, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.74 to 1.67] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Shared Decision Making - Feelings About Provider Involvement
Description: Patient report on 3-point scale of their feelings about provider involvement in contraceptive decision-making: I wish provider had been less involved, provider was involved the right amount, I wiss provider had been more involved.
Time Frame: Baseline (post-visit) and up to 24 months
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Right amount | 370 | 305
  Wish provider had been less involved | 8 | 10
  Wish provider had been more involved | 16 | 21
  Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who wished provider had been less involved to right amount (ref); Test type: Superiority; p = 0.85, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Relative risk ratio = 1.1, 95% CI 2-sided [0.40 to 3.04] — The estimation value represents the relative risk of the outcome in the intervention group, compared to relative risk in the control group
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who reported they wished their providers had been more involved, compared to right amount (ref); Test type: Superiority; p = 0.24, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Relative risk ratio = 1.6, 95% CI 2-sided [0.73 to 3.50] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Shared Decision Making - Provider Appropriately Expressed Preference
Description: Patient report of attitude on 3-point scale on how provider expressed preference for contraceptive method choice: Right amount, wish less strongly, wish more strongly.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  No, I wish less | 16 | 13
  Yes, exactly right | 357 | 297
  No, I wish more | 21 | 26
  Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who wished provider had expressed preference less strongly to right amount (ref); Test type: Superiority; p = 0.997, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Relative risk ratio = 1.00, 95% CI 2-sided [0.45 to 2.25] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who reported they wished provider had expressed preference more strongly, compared to right amount (ref); Test type: Superiority; p = 0.16, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Relative risk ratio = 0.69, 95% CI 2-sided [0.41 to 1.16] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Shared Decision Making - Satisfaction With How Provider Helped With Choice
Description: Patient report of satisfaction on a 5-point Likert scale (from 1=completely unsatisfied to 5=completely satisfied) of how the provider helped contraceptive method choice. Analyzed dichotomously as top score of 5 versus <5.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Completely satisfied | 303 | 240
  Less than completely satisfied | 91 | 96
  Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority — We ran a mixed effect regression model in a multiply imputed dataset, using fixed effects for study site and random effects for provider seen; p = 0.13, Regression, Logistic — P-value calculated in multiply imputed dataset; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.93 to 1.82] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Shared Decision Making - Who Made the Decision?
Description: Patient response to 5-point scale of who made decision on contraceptive method. The original 5 points were the provider by themselves, more provider, both equally, more patient, or provider by themselves. In analysis, these options were collapsed to three points: more provider, both equally, or more patient.
Time Frame: Baseline (post-visit)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Patient | 286 | 244
  Provider | 20 | 9
  Both | 88 | 83
  Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patient decision to both (ref); Test type: Superiority; p = 0.50, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Relative risk ratio = 1.13, 95% CI 2-sided [0.79 to 1.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of provider decision to both (ref); Test type: Superiority; p = 0.09, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Relative risk ratio = 2.14, 95% CI 2-sided [0.89 to 5.15] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Shared Decision Making - Provider Preference
Description: Patient report of whether or not provider had preference for contraceptive method choice, reported on a 5-point scale: no preference, slight preference, moderate preference, strong preference, extremely strong preference. Analyzed dichotomously as any preference versus no preference.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Provider had preference | 194 | 143
  Provider had no preference | 200 | 193
  Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p = 0.12, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.94 to 1.71] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Patient Decisional Conflict in Contraceptive Choice
Description: Patient Decisional Conflict was measured using the Decisional Conflict Scale (DCS), a validated measure to assess patients' decisional conflict in medical decision making. The DCS includes 16 items about experience of conflict, with 5-point Likert response options ranging from 0 ("Strongly disagree") to 4 ("Strongly agree"). Higher scores indicate less conflict. Top score on DCS (Range: 0-100, analyzed dichotomously as 100 versus <100). Top scores on subscales also analyzed (Informed decision, Uncertainty, Effective decision, Values clarity, Support, all ranging 0-100 and analyzed dichotomously as 100 versus <100).
Time Frame: Baseline (post-visit)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Overall score: Top score | 100 | 76
  Overall score: Less than top score | 294 | 260
  Overall score: Missing | 10 | 9
  Informed decision subscale: Top score | 199 | 145
  Informed decision subscale: Less than top score | 195 | 191
  Informed decision subscale: Missing | 10 | 9
  Uncertainty subscale: Top score | 164 | 112
  Uncertainty subscale: Less than top score | 230 | 224
  Uncertainty subscale: Missing | 10 | 9
  Effective decision subscale: Top score | 166 | 132
  Effective decision subscale: Less than top score | 228 | 204
  Effective decision subscale: Missing | 10 | 9
  Values clarity subscale: Top score | 196 | 154
  Values clarity subscale: Less than top score | 198 | 182
  Values clarity subscale: Missing | 10 | 9
  Support subscale: Top score | 207 | 172
  Support subscale: Less than top score | 187 | 164
  Support subscale: Missing | 10 | 9
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of overall score; Test type: Superiority; p = 0.41, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.80 to 1.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of informed decision subscale; Test type: Superiority; p = 0.0496, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.00 to 1.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of uncertainty subscale of DCS; Test type: Superiority; p = 0.03, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.03 to 2.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of effective decision subscale; Test type: Superiority; p = 0.5, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.80 to 1.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of values clarity subscale; Test type: Superiority; p = 0.31, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.86 to 1.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of support subscale; Test type: Superiority; p = 0.73, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.76 to 1.49] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Patient Knowledge of Contraceptive Options and Features
Description: Patient responses to items derived from National Survey of Reproductive Contraceptive Knowledge and previous studies of contraceptive knowledge and attitudes. All items analyzed as correct vs. incorrect.
Time Frame: Baseline (post-visit)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Pills are more effective than condoms: Correct | 220 | 170
  Pills are more effective than condoms: Incorrect | 174 | 166
  Pills are more effective than condoms: Missing | 10 | 9
  IUDs are more effective than pills: Correct | 279 | 162
  IUDs are more effective than pills: Incorrect | 115 | 174
  IUDs are more effective than pills: Missing | 10 | 9
  Depo is more effective than condoms: Correct | 238 | 156
  Depo is more effective than condoms: Incorrect | 156 | 180
  Depo is more effective than condoms: Missing | 10 | 9
  IUDs are an option for nulliparous young women: Correct | 315 | 228
  IUDs are an option for nulliparous young women: Incorrect | 79 | 108
  IUDs are an option for nulliparous young women: Missing | 10 | 9
  Methods causing periods to stop are safe: Correct | 305 | 220
  Methods causing periods to stop are safe: Incorrect | 89 | 116
  Methods causing periods to stop are safe: Missing | 10 | 9
  LARC can be removed early: Correct | 261 | 211
  LARC can be removed early: Incorrect | 133 | 125
  LARC can be removed early: Missing | 10 | 9
  Copper IUDs can act as EC: Correct | 89 | 33
  Copper IUDs can act as EC: Incorrect | 315 | 311
  Copper IUDs can act as EC: Missing | 0 | 1
  After sex, something to prevent pregnancy: Correct | 371 | 320
  After sex, something to prevent pregnancy: Incorrect | 23 | 16
  After sex, something to prevent pregnancy: Missing | 10 | 9
  EC can prevent pregnancy after sex: Correct | 361 | 315
  EC can prevent pregnancy after sex: Incorrect | 43 | 29
  EC can prevent pregnancy after sex: Missing | 0 | 1
  Pill does not affect fertility: Correct | 280 | 219
  Pill does not affect fertility: Incorrect | 114 | 117
  Pill does not affect fertility: Missing | 10 | 9
  Patch does not affect fertility: Correct | 277 | 201
  Patch does not affect fertility: Incorrect | 117 | 135
  Patch does not affect fertility: Missing | 10 | 9
  Ring does not affect fertility: Correct | 270 | 192
  Ring does not affect fertility: Incorrect | 124 | 144
  Ring does not affect fertility: Missing | 10 | 9
  Depo does affect fertility: Correct | 99 | 86
  Depo does affect fertility: Incorrect | 295 | 250
  Depo does affect fertility: Missing | 10 | 9
  Hormonal IUD does not affect fertility: Correct | 238 | 165
  Hormonal IUD does not affect fertility: Incorrect | 156 | 171
  Hormonal IUD does not affect fertility: Missing | 10 | 9
  Non-hormonal IUD does not affect fertility: Correct | 247 | 176
  Non-hormonal IUD does not affect fertility: Incorrect | 147 | 160
  Non-hormonal IUD does not affect fertility: Missing | 10 | 9
  Implant does not affect fertility: Correct | 233 | 164
  Implant does not affect fertility: Incorrect | 161 | 172
  Implant does not affect fertility: Missing | 10 | 9
  Composite IUD knowledge: Correct | 146 | 66
  Composite IUD knowledge: Incorrect | 258 | 279
  Composite IUD knowledge: Missing | 0 | 0
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - pills are more effective than condoms; Test type: Superiority; p = 0.12, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.94 to 1.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - IUDs are more effective than pills; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.65, 95% CI 2-sided [1.94 to 3.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - depo is more effective than condoms; Test type: Superiority; p = 0.0004, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.29 to 2.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - IUDs are an option for nulliparous young women; Test type: Superiority; p = 0.0002, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.36 to 2.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - Methods causing periods to stop are safe; Test type: Superiority; p = 0.001, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.28 to 2.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - LARC can be removed early; Test type: Superiority; p = 0.36, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.85 to 1.57] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of knowledge - Copper IUD can act as EC; Test type: Superiority; p < 0.0001, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.72 to 4.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of knowledge - After sex, there is something you can do to prevent pregnancy; Test type: Superiority; p = 0.49, Regression, Logistic — P-value calculated in multiply imputed dataset; We ran a regression model in a multiply imputed dataset. This outcome was not adjusted for site due to model being unable to run with imputed data; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.36 to 1.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of knowledge - EC can prevent pregnancy after sex; Test type: Superiority; p = 0.31, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 11, analysis 8]; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.39 to 1.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - pill does not affect fertility; Test type: Superiority; p = 0.08, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.96 to 1.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - patch does not affect fertility; Test type: Superiority; p = 0.002, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.2 to 2.26]; The odds ratio represents the odds of the intervention group in the numerator over the odds of the control group in the denominator
Statistical Analysis 12: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - ring does not affect fertility; Test type: Superiority; p = 0.002, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.23 to 2.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - Depo does affect fertility; Test type: Superiority; p = 0.77, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.62 to 1.43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - Hormonal IUD does not affect fertility; Test type: Superiority; p = 0.002, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.19 to 2.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - Non-hormonal IUD does not affect fertility; Test type: Superiority; p = 0.004, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.15 to 2.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - Implant does not affect fertility; Test type: Superiority; p = 0.005, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.14 to 2.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of correct knowledge - composite IUD knowledge item (all correct responses on items related to IUD knowledge, versus any incorrect); Test type: Superiority; p < 0.0001, Regression, Logistic — P-value calculated in multiply imputed dataset; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.75 to 3.49] — OR calculated in multiply imputed dataset. Intervention patients had 2.47 times the odds of control patients to give correct answer

12. Secondary Outcome: Patient Chosen Contraceptive Method Satisfaction
Description: 5-point Likert scale item regarding patient satisfaction with contraceptive method chosen at baseline visit. The item is a statement of method satisfaction, and response options range from 1 ("Completely disagree") to 5 ("Completely agree"). A higher score indicates higher satisfaction. Analyzed dichotomously as top score (5) versus all lower scores.
Time Frame: Reported and analyzed at baseline (post-visit), 4 months and 7 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Baseline: Top score of 5 | 249 | 199
  Baseline: Less than top score | 145 | 137
  Baseline: Missing | 10 | 9
  4 months post-enrollment: Top score of 5 | 176 | 157
  4 months post-enrollment: Less than top score | 183 | 148
  4 months post-enrollment: Missing | 45 | 40
  7 months post-enrollment: Top score of 5 | 180 | 160
  7 months post-enrollment: Less than top score | 177 | 130
  7 months post-enrollment: Missing | 47 | 55
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of percentage of patients giving top score at baseline; Test type: Superiority; p = 0.25, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.88 to 1.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of percentage of patients giving top score at 4 months post-enrollment; Test type: Superiority; p = 0.5, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.66 to 1.22] — The odds ratio represents the odds of the intervention groups in the numerator over the odds of the control group in the denominator
Statistical Analysis 3: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of percentage of patients giving a top score on the 5-point Likert scale at 7 months post-enrollment; Test type: Superiority; p = 0.23, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.60 to 1.13] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Patient Current Contraceptive Method Satisfaction
Description: 5-point Likert scale question regarding patient satisfaction with the contraceptive method they are currently using. The item is a statement of method satisfaction, and response options range from 1 ("Completely disagree") to 5 ("Completely agree"). A higher score indicates higher satisfaction. Analyzed dichotomously as top score of 5 versus <5.
Time Frame: 7 months follow-up
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Completely satisfied | 209 | 177
  Less than completely satisfied | 147 | 113
  Missing | 48 | 55
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p = 0.55, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.66 to 1.25] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Patient Attitude Towards Use of Contraceptive Options
Description: Patient ratings of contraceptive methods on the 11-point Global Contraceptive Attitude scale, developed by the PI. To assess overall (or "global") attitude towards use of various methods, patients are asked to respond the following with regard to each method listed in the data table: "Overall, how would you rate each of the following as a birth control method for yourself, (even if you've never used it)?" Response options range from 0 ("Terrible method") to 10 ("Great method"). A higher score on an individual item indicates a more positive attitude towards a method. Analyzed as discrete items with responses of 0 to 10; item scores not combined into an overall scale score.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Units on a scale
  Pill | 6.26 (0.24) | 6.55 (.289)
  Patch | 5.22 (0.20) | 5.4 (0.19)
  Ring | 5.07 (0.18) | 5.49 (0.26)
  Shot | 5.05 (0.18) | 5.35 (0.19)
  Hormonal IUD | 6.61 (.23) | 6.24 (.18)
  Non-hormonal IUD | 6.3 (0.21) | 6.29 (0.17)
  Implant | 5.79 (0.16) | 6.06 (0.20)
  Condoms | 6.33 (0.16) | 6.87 (0.15)
  Withdrawal | 2.8 (0.15) | 2.98 (0.21)
  Female sterilization | 4.44 (0.27) | 5.59 (0.24)
  Male sterilization | 4.98 (0.25) | 6.08 (0.28)
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating for hormonal IUD. Patients excluded from analysis if they had not heard of hormonal IUD; Test type: Superiority; p = 0.13, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.92 to 1.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on non-hormonal IUD. Patients were excluded from this analysis if they reported not having heard of the non-hormonal IUD in the post-visit survey; Test type: Superiority; p = 0.92, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.75 to 1.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Contraceptive Decision Support Tool; Comparison of rating of implant; Test type: Superiority; p = 0.17, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.67 to 1.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on condoms. Patients were excluded from this analysis if they reported not having heard of condoms in the post-visit survey; Test type: Superiority; p = 0.009, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.54 to 0.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on the shot (Depo Provera). Patients were excluded from this analysis if they reported not having heard of the the shot (Depo Provera) in the post-visit survey; Test type: Superiority; p = 0.26, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.65 to 1.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on the pill. Patients were excluded from this analysis if they reported not having heard of the pill in the post-visit survey; Test type: Superiority; p = 0.23, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.64 to 1.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on the patch. Patients were excluded from this analysis if they reported not having heard of the patch in the post-visit survey; Test type: Superiority; p = 0.55, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.69 to 1.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on the pull-out method. Patients were excluded from this analysis if they reported not having heard of the pull-out method in the post-visit survey; Test type: Superiority; p = 0.84, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.76 to 1.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on the ring. Patients were excluded from this analysis if they reported not having heard of the ring in the post-visit survey; Test type: Superiority; p = 0.07, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.64 to 1.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on female sterilization/tubal ligation. Patients were excluded from this analysis if they reported not having heard of female sterilization/tubal ligation in the post-visit survey; Test type: Superiority; p = 0.002, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.42 to 0.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of rating on male sterilization/vasectomy. Patients were excluded from this analysis if they reported not having heard of male sterilization/vasectomy in the post-visit survey; Test type: Superiority; p = 0.005, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.4 to 0.85] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Newly Heard About Methods During Visit
Description: Percentage of patients who reported having heard about a method in the post-survey, but not the pre-survey.
Time Frame: Baseline (pre- and post-survey)
Population: Only calculated for those patients who reported not having heard of method in pre-survey, and then completed post-survey. All other patients missing for this item and excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Newly heard of hormonal IUD: Yes | 79 | 46
  Newly heard of hormonal IUD: No | 21 | 18
  Newly heard of hormonal IUD: Missing | 304 | 281
  Newly heard of non-hormonal IUD: Yes | 104 | 84
  Newly heard of non-hormonal IUD: No | 23 | 31
  Newly heard of non-hormonal IUD: Missing | 277 | 230
  Newly heard of implant: Yes | 80 | 58
  Newly heard of implant: No | 30 | 26
  Newly heard of implant: Missing | 294 | 261
  Newly heard of patch: Yes | 39 | 38
  Newly heard of patch: No | 11 | 19
  Newly heard of patch: Missing | 354 | 288
  Newly heard of ring: Yes | 61 | 41
  Newly heard of ring: No | 24 | 23
  Newly heard of ring: Missing | 319 | 281
  Newly heard of male sterilization: Yes | 53 | 35
  Newly heard of male sterilization: No | 30 | 24
  Newly heard of male sterilization: Missing | 321 | 286
  Newly heard of female sterilization: Yes | 59 | 44
  Newly heard of female sterilization: No | 27 | 26
  Newly heard of female sterilization: Missing | 318 | 275
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of hormonal IUD; Test type: Superiority; p = 0.27, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.71 to 3.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of non-hormonal IUD; Test type: Superiority; p = 0.18, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.80 to 3.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of implant; Test type: Superiority; p = 0.5, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.62 to 2.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of the patch; Test type: Superiority; p = 0.32, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.59 to 4.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of ring; Test type: Superiority; p = 0.37, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.68 to 2.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of male sterilization (vasectomy); Test type: Superiority; p = 0.39, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.60 to 3.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison of patients who newly heard of female sterilization; Test type: Superiority; p = 0.39, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.6 to 3.73] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Patient Rating of Visit as "Much Better" Than Previous Family Planning Visit
Description: Patient report on 5-point Likert scale question asking patient to compare this visit to last family planning visit (1=Today was much worse; 5=today was much better). Analyzed dichotomously as top score of 5 versus <5.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only. Only calculated among those participants who reported ever having had a family planning visit. All others missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Much better | 142 | 104
  Not much better | 144 | 140
  Missing | 118 | 101
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Patients excluded from test if they reported not having had a previous contraceptive counseling appointment; Test type: Superiority; p = 0.18, Regression, Logistic — P-value calculated from multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.90 to 1.81] — The odds ratio represents the odds of the intervention group rating their appointment as "much better," in the numerator, over the odds of the control group giving this rating in the denominator

17. Secondary Outcome: Total Clinic Visit Time
Description: Total amount of time a patient spends in a clinic for a family planning visit, from check-in to check-out.
Time Frame: Baseline visit
Population: Observed in patients only
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
minutes | 98.40 (1.75) | 86.94 (1.71)
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p < 0.001, Regression, Linear — P-value calculated in multiple imputed dataset; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 11.81, 95% CI 2-sided [8.54 to 18.66] — The estimation parameter is a beta coefficient from a linear regression model, calculated in an imputed dataset. It represents additional minutes in an intervention visit versus a control visit

18. Secondary Outcome: Time Spent With Contraceptive Counseling Provider
Description: Total amount of time spent with the provider that is providing contraceptive counseling.
Time Frame: Baseline visit
Population: Observed in patients
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
minutes | 44.0 (1.21) | 44.4 (1.29)
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p = 0.63, Regression, Linear — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [-3.19 to 5.29] — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: Maslach Burnout Inventory
Description: Provider participants were asked to respond to the Maslach Burnout Inventory on workplace burnout among human services workers. The scale includes 22 items with response options on a Likert scale of 0-6. Individual scores were calculated at both baseline and follow-up for three subscales: emotional exhaustion (Range: 0-54, with higher score representing higher emotional exhaustion), depersonalization (Range: 0-30, with a higher score representing higher depersonalization), and personal accomplishment (Range: 0-48, with a higher score representing more personal accomplishment in the workplace).
Time Frame: Change between baseline and end of study (up to 24 months post-enrollment). In multivariate analysis, follow-up score analyzed controlling for site and score at baseline (Analyses 1-3).
Population: Observed in providers only
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Contraceptive Decision Support Tool Providers: Providers randomized to use the contraceptive decision support tool and to use to the tool with their patients participating in the study.
- Usual Care Providers: Providers randomized to practice usual care with their patients participating in the study.
Arm/Group | Contraceptive Decision Support Tool Providers | Usual Care Providers
Number analyzed (Participants) | 15 | 13
Units on a scale
  Change in emotional exhaustion | -2.27 (9.22) | 1.07 (9.38)
  Change in depersonalization | -0.87 (4.10) | 0.46 (4.24)
  Change in personal accomplishment | -0.80 (3.99) | 2.38 (5.30)
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool Providers vs Usual Care Providers; Test of follow-up score of emotional exhaustion subscale of Maslach Burnout Inventory, controlling for baseline score and site; Test type: Superiority; p = 0.24, Regression, Linear; Observed coefficient = -3.97, 95% CI 2-sided [-10.62 to 2.68], Standard Error of Mean 3.34 — Tool group is compared to control group (ref). Bootstrapping used for standard error
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool Providers vs Usual Care Providers; Linear regression of follow-up score for depersonalization subscale of Maslach Burnout Inventory, controlling for baseline score and site; Test type: Superiority; p = 0.36, Regression, Linear; Observed coefficient = -1.52, 95% CI 2-sided [-4.76 to 1.72], Standard Error of Mean 1.91 — Tool group is compared to control group (ref). Bootstrapping used for standard error
Statistical Analysis 3: Comparison: Contraceptive Decision Support Tool Providers vs Usual Care Providers; Linear regression of follow-up score for personal accomplishment subscale of Maslach Burnout Inventory, controlling for site and baseline score; Test type: Superiority; p = 0.28, Regression, Linear; Slope = -1.64, 95% CI 2-sided [-4.61 to 1.34], Standard Error of Mean 1.34 — Tool group compared to control group (ref). Bootstrapping used for standard error

20. Other Pre Specified Outcome: Choice of a Highly Effective Method of Contraception at Baseline
Description: Patient report of whether or not patient chose highly effective method at baseline. Highly effective methods include implants, IUDs, and male and female sterilization.
Time Frame: Baseline (post-visit survey)
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  Chose highly effective method | 153 | 120
  Did not choose highly effective method | 249 | 221
  Missing | 2 | 4
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Test type: Superiority; p = 0.78, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.69 to 1.65] — [estimate comment as in outcome 1, analysis 1]

21. Other Pre Specified Outcome: Use of a Highly Effective Method of Contraception at 4 and 7 Months Follow-up.
Description: Whether patient is using a highly effective contraceptive method at 4 and 7 month follow-up survey. Highly effective methods include implant, IUDs, and male and female sterilization.
Time Frame: 4 and 7 months post-enrollment
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  At 4 months: Yes | 264 | 230
  At 4 months: No | 94 | 76
  At 4 months: Missing | 46 | 39
  At 7 months: Yes | 258 | 201
  At 7 months: No | 99 | 90
  At 7 months: Missing | 47 | 54
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 4 months post-enrollment; Test type: Superiority; p = 0.75, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.66 to 1.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 7 months post-enrollment; Test type: Superiority; p = 0.71, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.75 to 1.53] — [estimate comment as in outcome 1, analysis 1]

22. Other Pre Specified Outcome: Use of Any Moderately or Highly Effective Method of Contraception at 4 and 7 Months Follow-up
Description: Patient report of whether or not patient is using a highly or moderately effective contraceptive method at 4 and 7 month follow-up survey. As defined by the Centers for Disease Control, moderately effective methods include injectables, pills, patch, vaginal ring, and diaphragm; typical failure rates range from 6-12%. Highly effective methods include implants, IUDs, and male and female sterilization; failure rates are less than 1%.
Time Frame: 4 and 7 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  At 4 months post-enrollment: Yes | 264 | 230
  At 4 months post-enrollment: No | 94 | 76
  At 4 months post-enrollment: Missing | 46 | 39
  At 7 months post-enrollment: Yes | 258 | 201
  At 7 months post-enrollment: No | 99 | 90
  At 7 months post-enrollment: Missing | 47 | 54
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 4 months post-enrollment; Test type: Superiority; p = 0.75, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.66 to 1.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 7 months post-enrollment; Test type: Superiority; p = 0.37, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.83 to 1.64] — [estimate comment as in outcome 1, analysis 1]

23. Other Pre Specified Outcome: Unplanned Pregnancy
Description: Incidence of unplanned pregnancy among study participants, as determined by responses of patients who experienced a pregnancy to the 6-item London Measure of Unplanned Pregnancy. The London Measure includes items on attitude towards an experienced pregnancy and behaviors before pregnancy to determine the intendedness of pregnancy. The score range of the London Measure is 0-12, with a score of <10 indicating unplanned pregnancy and a score of 10 or higher indicating planned pregnancy. We report the percentage of patients who report a pregnancy and report a score of <10 on the London Measure.
Time Frame: 4 months and 7 months from enrollment
Population: Observed in patients only
Measure: Count of Participants; unit: Participants
Arm/Group | Contraceptive Decision Support Tool | Usual Care (Control)
Number analyzed (Participants) | 404 | 345
Participants
  At 4 months post-enrollment: Yes | 11 | 8
  At 4 months post-enrollment: No | 350 | 300
  At 4 months post-enrollment: Missing | 43 | 37
  At 7 months post-enrollment: Yes | 24 | 11
  At 7 months post-enrollment: No | 336 | 280
  At 7 months post-enrollment: Missing | 44 | 54
Statistical Analysis 1: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 4 months post-enrollment; Test type: Superiority; p = 0.63, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.48 to 3.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Contraceptive Decision Support Tool vs Usual Care (Control); Comparison at 7 months post-enrollment; Test type: Superiority; p = 0.11, Regression, Logistic — P-value calculated in multiply imputed dataset; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.88 to 3.80] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 7 months (from patient enrollment through study period)
Groups:
- Contraceptive Decision Support Tool Providers: Providers randomized to use the tool with their study patients.
- Usual Care (Control) Providers: Providers randomized to deliver usual care to their study patients.
Arm/Group | Contraceptive Decision Support Tool Patients | Usual Care (Control) Patients | Contraceptive Decision Support Tool Providers | Usual Care (Control) Providers
All-Cause Mortality (participants affected / at risk) | 0/407 | 0/351 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/407 | 0/351 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/407 | 0/351 | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Limitations include potential for contamination between provider arms, our inability to blind patients or providers due to the nature of the intervention, and the potential for unobserved differences between patient arms due to cluster randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02078713/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT02078713/SAP_001.pdf